CLINICAL TRIAL: NCT01802996
Title: A Randomized, Controlled, Multi-center Collaborative Study to Evaluate the Efficacy of Magnesium Isoglycyrrhizinate Injection in the Prevention of Antineoplastic Chemotherapy Related Acute Liver Injury
Brief Title: Evaluate the Efficacy of Magnesium Isoglycyrrhizinate in the Prevention of Chemotherapy Related Acute Liver Injury
Acronym: MAGIC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cttq (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MAGIC-301
Record Dates: First submitted 2013-02-26; First posted 2013-03-04 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Neoplasms; Liver Injury
MeSH Terms: conditions — Neoplasms | interventions — 18alpha,20beta-hydroxy-11-oxo-norolean-12-en-3beta-yl-2-O-beta-D-glucopyranurosyl-alpha-D-glucopyranosiduronate magnesium tetrahydrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Magnesium Isoglycyrrhizinate Injection 200mg IV on days 1-5
  Interventions: Drug: Magnesium Isoglycyrrhizinate Injection
- Arm II (No Intervention): Only chemotherapy

INTERVENTIONS:
Drug: Magnesium Isoglycyrrhizinate Injection — 200mg IV on day 1-5
  Other Names: Tianqingganmei®; 2005S07127
  Arms: Arm I

SUMMARY:
This purpose of this study is to evaluate the evaluate the efficacy of Magnesium Isoglycyrrhizinate Injection in the prevention of antineoplastic chemotherapy related acute liver injury.

DETAILED DESCRIPTION:
Total subjects: 2040, experimental group of 1360 patients, control group of 680 patients. According to the study subjects receiving antineoplastic chemotherapy, subjects are stratified randomize.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-75 years;
2. Patients with malignant tumor accord with chemotherapy indication, candidate to a chemotherapy treatment, disease is not restricted;
3. Accorded with the following chemotherapy plan: included cis-platinum, ≥60mg/m2/course; included oxaliplatin, ≥85mg/m2/course; included cyclophosphamide, ≥600mg/m2/course; included gemcitabine, ≥60mg/m2/course;
4. ECOG≤2;
5. Estimates survival time≥3 months;
6. TBIL≤1.0×ULN, ALT、AST≤1.0×ULN; blood examination, uronoscopy, stool examination, renal function tests and electrocardiogram are normal;
7. Patients have been apart from the previous chemotherapy to finish above 2 weeks (including 2 weeks).

Exclusion Criteria:

1. Patients with partial liver radiotherapy;
2. Hepatitis B or C virus replication in the state, the patient will need antiviral therapy;
3. Patients have serious heart diseases, liver kidney diseases, or metabolism function disorder;
4. Patients combined with cellular immune therapy;
5. Within 2 weeks of application or currently possible applications of drugs(polyene phosphatidylcholine, reduced glutathione, tiopronin and other hepatoprotective and choleretic drugs), interference with the study;
6. Pregnancy, or patients during breast feeding;
7. Patients have known hypersensitivity to Glycyrrhizin;
8. Patients are participating, or have participated in other Clinical studies of new drugs within 4 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2040 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
The incidence of liver injury | 0-15 days
  anyone of ALT、AST、ALP、TBIL、DBIL、γ-GT>ULN

CONTACTS AND LOCATIONS:
Overall Officials: Qin Shukui, MD, Principal Investigator — The 81st hospital of PLA
Locations (27):
- China (27):
  - The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine, Hefei, Anhui
  - China PLA General Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of General Hospital of PLA ( 304 ), Beijing, Beijing Municipality
  - Fujian Province-owned Hospital, Fuzhou, Fujian
  - Fuzhou General Hospital of Nanjing Military Area Command, Fuzhou, Fujian
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong
  - Tumour Hospital Affiliated to Guangzhou Medical College, Guangzhou, Guangdong
  - The Affiliated Tumor Hospital of Guangxi Medical University, Nanning, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The first hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The second hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The people's Hospital of Wuhan University, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Changzhou Second People's Hospital, Changzhou, Jiangsu
  - The 81st hospital of PLA, Nanjing, Jiangsu
  - Nanjing General Hospital of Nanjing Military Area Command, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The first hospital of Nanjing, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Wuxi Fourth People's Hospital, Wuxi, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Affiliated Hospital of Medical College of Qiingdao University, Qingdao, Shandong
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang